CLINICAL TRIAL: NCT04326244
Title: The Relationship Between Obesity-related Molecular Typing and Traditional Chinese Medicine Constitution
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG1H0052
Record Dates: First submitted 2020-03-09; First posted 2020-03-30 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-02

CONDITIONS: Obstructive Sleep Apnea; Obesity
Keywords: Obesity; Obstructive Sleep Apnea; Gene; Traditional Chinese medicine constitution
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Hematologic Tests; Genetic Testing; Cephalometry; Polysomnography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Snoring obesity patient: Constitution in Chinese Medicine Questionnaire, physical examination, blood test and genetic test are provided to subjects. The blood test includes High-density lipoprotein- cholesterol, Low-density lipoprotein- cholesterol, Total cholesterol, Triglyceride, Leptin, Glucose AC, Hemoglobin A1C, Insulin; the DNA test includes FTO、MC4R、BDNF、PPARG、ADRB3、UCP1. Epworth Sleepiness Scale, laryngoscope and polysomnography are also performed in the patients enrolled
  Interventions: Diagnostic Test: blood test; Diagnostic Test: genetic test; Diagnostic Test: Constitution in Chinese Medicine Questionnaire; Diagnostic Test: Epworth Sleepiness Scale; Diagnostic Test: cephalometry; Diagnostic Test: polysomnography

INTERVENTIONS:
Diagnostic Test: blood test — High-density lipoprotein- cholesterol, Low-density lipoprotein- cholesterol, Total cholesterol, Triglyceride, Leptin, Glucose AC, Hemoglobin A1C, Insulin
Diagnostic Test: genetic test — FTO、MC4R、BDNF、PPARG、ADRB3、UCP1
Diagnostic Test: Constitution in Chinese Medicine Questionnaire — Constitution in Chinese Medicine Questionnaire
Diagnostic Test: Epworth Sleepiness Scale — Epworth Sleepiness Scale
Diagnostic Test: cephalometry — Evaluation of craniofacial morphology in OSA patients
Diagnostic Test: polysomnography — to evaluate Apnea-Hypopnea Index (AHI) for the severity of sleep apnea

SUMMARY:
Obesity is an epidemic and a growing problem in the world. There are numerous causes of obesity, the most novel and personalized of which is genetic inheritance. Single nucleotide polymorphisms are the most common type of genetic variation among people, regulating the response between the diet and the body. Meanwhile, Traditional Chinese medicine pattern differentiation is also personalized and usually influenced by inheritance, living habits, character and environment and so on. The common constitutions in obesity are Qi deficiency, Yang Deficiency, and Phlegm dampness, which are correlated with oxygen, sugar and fat metabolism, also affected by gene expression. Therefore, the relationship between constitution, metabolism and genetic molecular typing may be significant in obesity with obstructive sleep apnea patients.

DETAILED DESCRIPTION:
Method The adults whose age between 20~65 years old, BMI between 27kg/m² and 35kg/m², and also have snoring during sleeping are able to be enrolled in the study. Then, the general data questionnaire, Body Constitution Questionnaire, physical examination, blood test, and genetic test are provided to subjects. The blood test includes High-density lipoprotein- cholesterol, Low-density lipoprotein- cholesterol, Total cholesterol, Triglyceride, Leptin, Glucose AC, Hemoglobin A1C, Insulin; the DNA test includes FTO、MC4R、BDNF、PPARG、ADRB3、UCP1. Epworth Sleepiness Scale, laryngoscope and polysomnography are also performed in the patients enrolled. The Traditional Chinese medicine constitution can be classified and its relationship between different figure types, serum lipid level as well as obesity-related gene can be analyzed. The results will be described after a statistical analysis.

Aim The aim of this study is to analyze the constitution, finding the association between obesity patients with obstructive sleep apnea and their related molecular typing and Traditional Chinese Medicine constitution.

ELIGIBILITY:
Inclusion Criteria:

1. 27≦BMI≦35 kg/m² and with snoring during sleeping
2. 20y/o<age<65y/o with conscious clear
3. no recognition impairment
4. could accept blood test and questionnaire
5. willing to sign Informed consent

Exclusion Criteria:

1. age<20 years old
2. pregnancy or women under breastfeeding
3. patients have been diagnosed with endocrine disorders such as thyroid, adrenal and autoimmune disease
4. patients have been diagnosed with neurological or psychological disorders with recognition impairment
5. Patients with severe visual, hearing, or physical impairment that would interfere with questionnaire processing.
6. Patients are under other experimental medication
7. Patients are under weight-loss drug in recent one month

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obesity patient with Obstructive sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Obesity-related gene profile | At enrollment
  Examine Obesity-related gene profile: FTO, MC4R, BDNF, PPARG, ADRB3, UCP1 to evaluate the association between gene profile and obstructive sleep apnea (OSA) or traditional Chinese medicine (TCM) constitution.
Constitution in Chinese Medicine Questionnaire | At enrollment
  The scale classification of the patient's constitution according to Traditional Chinese Medicine theory into nine constitutions. The Constitution in Chinese Medicine Questionnaire (CCMQ) consists of 60 items to classify a person into one or more of nine body constitution types: balanced (8 Items), Qi-deficiency (8 Items), Yang-deficiency (7 Items), Yin-deficiency (8 Items), phlegm-wetness (8 Items), wetness-heat (6 Items), blood-stasis (7 Items), Qi-depression (7 Items), and special diathesis (7 Items). A higher score in the CCMQ scale indicates a higher likelihood of the specific body constitution. The original score is sum up each item's score. The converted scores is [(original scores- items)/(items*40]*100. The balanced constitution is the converted score >60 and the rest constitutions' converted scores all < 30. The unbalanced constitution is the converted score ≥40.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | At enrollment
  The severity evaluation of impact on lethargy caused by obstructive sleep apnea. The total score can range from 0 to 24. A higher score is associated with increased sleepiness.
Polysomnography | At enrollment
  The evaluation on obstructive sleep apnea severity
Cephalometry | At enrollment
  The evaluation on cranial morphology of enrolled patients
Lipid profile (mg/dl) | At enrollment
  Includes High-density lipoprotein- cholesterol, Low-density lipoprotein- cholesterol, Total cholesterol, Triglyceride.
Serum leptin test (ng/mL) | At enrollment
  High serum leptin level is related to obesity
Glucose AC (mg/dL) | At enrollment
  High glucose AC is related to diabetes.
HbA1C (Glycohemoglobin, %) | At enrollment
  High HbA1C is related to diabetes.
Insulin (uU/mL) | At enrollment
  HOMA-IR index (Homeostasis Model Assessment-Insulin Resistance index) is calculated by Insulin with Glucose AC to evaluate the insulin resistance of enrolled patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Hao Jiang, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bielicki P, Plywaczewski R, Brzoska K, Kumor M, Barnas M, Jonczak L, Stepkowski TM, Piechuta A, Chazan R, Sliwinski P, Kruszewski M. Impact of polymorphism of selected genes on the diagnosis of type 2 diabetes in patients with obstructive sleep apnea. Pol Arch Intern Med. 2019 Jan 31;129(1):6-11. doi: 10.20452/pamw.4406. Epub 2018 Dec 29. PMID 30600310
- [Background] Shah F, Forsgren S, Holmlund T, Levring Jaghagen E, Berggren D, Franklin KA, Stal P. Neurotrophic factor BDNF is upregulated in soft palate muscles of snorers and sleep apnea patients. Laryngoscope Investig Otolaryngol. 2018 Nov 28;4(1):174-180. doi: 10.1002/lio2.225. eCollection 2019 Feb. PMID 30828636
- [Background] Jiao X, Yang S, Yang Y, Li J, Sun H, Zhang M, Yang Y, Qin Y. Targeted sequencing analysis of PPARG identifies a risk variant associated with obstructive sleep apnea in Chinese Han subjects. Sleep Breath. 2020 Mar;24(1):167-174. doi: 10.1007/s11325-019-01855-x. Epub 2019 May 2. PMID 31044373
- [Background] Pierola J, Barcelo A, de la Pena M, Barbe F, Soriano JB, Sanchez Armengol A, Martinez C, Agusti A. beta3-Adrenergic receptor Trp64Arg polymorphism and increased body mass index in sleep apnoea. Eur Respir J. 2007 Oct;30(4):743-7. doi: 10.1183/09031936.00152006. Epub 2007 Jul 11. PMID 17626108
- [Background] Thorleifsson G, Walters GB, Gudbjartsson DF, Steinthorsdottir V, Sulem P, Helgadottir A, Styrkarsdottir U, Gretarsdottir S, Thorlacius S, Jonsdottir I, Jonsdottir T, Olafsdottir EJ, Olafsdottir GH, Jonsson T, Jonsson F, Borch-Johnsen K, Hansen T, Andersen G, Jorgensen T, Lauritzen T, Aben KK, Verbeek AL, Roeleveld N, Kampman E, Yanek LR, Becker LC, Tryggvadottir L, Rafnar T, Becker DM, Gulcher J, Kiemeney LA, Pedersen O, Kong A, Thorsteinsdottir U, Stefansson K. Genome-wide association yields new sequence variants at seven loci that associate with measures of obesity. Nat Genet. 2009 Jan;41(1):18-24. doi: 10.1038/ng.274. Epub 2008 Dec 14. PMID 19079260
- [Background] Yeo GSH. Genetics of obesity: can an old dog teach us new tricks? Diabetologia. 2017 May;60(5):778-783. doi: 10.1007/s00125-016-4187-x. Epub 2016 Dec 24. PMID 28013339
- [Background] Yang Q, Xiao T, Guo J, Su Z. Complex Relationship between Obesity and the Fat Mass and Obesity Locus. Int J Biol Sci. 2017 May 15;13(5):615-629. doi: 10.7150/ijbs.17051. eCollection 2017. PMID 28539834